CLINICAL TRIAL: NCT02870088
Title: The Effect of Breaking Prolonged Sitting on Adipose Tissue and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Ministry of Education, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yung-Chih Chen, PhD student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13/SW/0321
Record Dates: First submitted 2016-02-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Sitting (Active Comparator): Participants sat on a chair during the trial.
  Interventions: Behavioral: Prolonged Sitting
- Breaking Sitting (Experimental): Participants walked regularly during the trial.
  Interventions: Behavioral: Breaking Sitting

INTERVENTIONS:
Behavioral: Prolonged Sitting — After consuming 1st meal, participants sat on a chair for 180 min. After 180 min, the 2nd meal was provided. After finishing the 2nd meal, participants sat on a chair for another 120 min.
  Arms: Prolonged Sitting
Behavioral: Breaking Sitting — After consuming 1st meal, participants walked 2 min on a treadmill every 20 minutes for the following 180 min. For the remainder of the time participants sat on the chair. After 180 min, the 2nd meal was provided. After finishing the 2nd meal, participants continued 2 min of walking every 20 min for the following 120 min.
  Arms: Breaking Sitting

SUMMARY:
The purpose of this project is to investigate the effect of breaking prolonged sitting on acute adipose tissue and metabolic responses.

DETAILED DESCRIPTION:
Pre-trial assessments:

Physical activity assessment : a combined heart rate/accelerometer monitor was worn for 7 days to assess participant's habitual physical activity energy expenditure (Actiheart, Cambridge Neurotechnology Ltd., Cambridge, UK). This was attached to the left chest via 2 adhesive ECG pads for 24 hours per day except for during showering/bathing/swimming.

Body composition analysis:

Body mass was assessed using digital scales post-void (TANITA corp., Tokyo, Japan). Waist and hip circumference was assessed based on World Health Organisation guidelines. Body composition was determined by using Dual energy X-ray absorptiometry (Discovery, Hologic, Bedford, UK). Abdominal subcutaneous and visceral adipose tissue mass was estimated from a central region between L1-L4.

Trial days:

In the 72 h prior to each main trial, participants were asked to refrain from performing any strenuous physical activity. In the 48 h prior to each main trial, consuming alcohol/caffeine was not allowed and in the meantime, a dietary record was completed 48 h before the first main trial. Participants were asked to replicate this diet prior to their second main trial. In addition, in the 48 h prior to each main trial, participants were asked to restrict their steps to under 4000 steps per day in order to mimic sedentary lifestyle patterns and eliminate any acute effects from recent physical activity.

Two trials were performed including one prolonged sitting and one breaking prolonged sitting trials. In the breaking trial, after consuming 1st meal, participants walked 2 min on a treadmill at 6.4 km/h speed every 20 minutes for the following 180 min. For the remainder of the time participants sat on the chair. After 180 min, the 2nd meal was provided. After finishing the 2nd meal, participants were continue 2 min of breaking prolonged sitting physical activity at the same speed every 20 min for the following 120 min. In total, participants performed 15 two minute bouts of physical activity throughout the trial for a total of 30 min breaking prolonged sitting physical activity. In the prolonged sitting trial, participants sat on a chair.

Expired air, RPE and heart rate were collected in two of breaking sitting walks to determine exercise intensity and energy expenditure. In addition, two 5 min sitting of expired air and heart rate were taken to calculated total energy expenditure during sitting. During each trial, participants were allowed to move from a sitting position to the treadmill or to void if required. While sitting, participants were only allowed to read, use a laptop or watch television but were otherwise asked to keep as still as possible throughout. In the first trial, participants were allowed to consume water ad libitum and the volume ingested was replicated for the 2nd trial

In each main trial, baseline blood samples was collected before the 1st meal and hourly for the following 5 hours. Additional blood samples were collected every 15 min after the first and second meal. A total of 14 blood samples were collected for each trial.

Adipose tissue culture and gene expression:

After adipose tissue biopsy and cleaning, tissue was minced to approximately 5-10 mg and directly placed in sterile culture plates (Nunc, Roskilde, Denmark) with endothelial cell basal media (ECBM) containing 0.1% fatty acid-free bovine serum albumin 100 U ml-1 penicillin and 0.1 mg ml-1 streptomycin (Sigma-Aldrich, Gillingham, UK). Adipose tissue was incubated with a final ratio of 100mg tissue per 1 ml ECBM media for 3 hours. A 37°C, 5% CO2 and 95 ± 5% relative humidity incubator was used (MCO-18A1C CO2 incubator; Sanyo, Osaka, Japan). Media was transferred to sterile eppendorfs and stored at -80°C after 3 hours incubation. Approximately 200 mg adipose tissue was homogenised in 5ml Trizol in an RNase/DNase-free sterile tube (Invitrogen, Paisley, UK) and stored at -80°C before further analysis.

Sample size:

A previous similar study reported incremental area under curve (iAUC) for insulin during breaking prolonged sitting compared to prolonged sitting of 3337 IU L-1 9h-1 and 2470 IU L-1 9h-1, respectively. Based on an assumed SD of 600 IU L-1 9h-1, we would require 9 participants to show a difference in iAUC for insulin with 95% power and 5% alpha.

Statistics:

All data was presented as mean ± standard error of mean (SEM). Incremental area under curve (iAUC) was calculated using the trapezoid method and differences between trials analysed using paired t-tests. Glucose, insulin, NEFA, adipokines, and cell culture outcomes were determined using a two-way ANOVA with repeated measures using SPSS version 22 (IBM, Armonk, NY, USA). Where significant interactions (trial × time) were found, a post hoc analysis was applied using t-test with the Holm-Bonferroni correction. Single comparisons used a t-test or non-parametric equivalent. Statistical significance was set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and post-menopausal females (post-menopausal diagnosis based on consecutive absence of menstrual cycles for >12 months).
* Aged between 35 and 64 years
* Central overweight (waist circumference greater than 94 cm for males and 80 cm for females)
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker
* Able to walk comfortably on a treadmill

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Waist circumference < 94cm for male and < 80cm for female
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function
* Unable to take part in exercise for any reason (e.g., injury or disability) or a positive response to any questions on the Physical Activity Readiness questionnaire (PAR-Q)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incremental area under curve (iAUC) for insulin | 330 minutes

SECONDARY OUTCOMES:
Changes in gene expression in the adipose tissue | Before the 1st meal and 120 min after the 2nd meal (330 minutes).
Changes in insulin, glucose, TAG and NEFA in blood | 330 minutes
Changes in serum Interleukin-6 (IL-6), leptin and adiponectin | 330 minutes
Changes in Interleukin-6 (IL-6), leptin and adiponectin protein secretion from adipose tissue explants | Before the 1st meal and 120 min after the 2nd meal (330 minutes).

IPD SHARING:
Plan to Share IPD: Undecided